CLINICAL TRIAL: NCT02516488
Title: Comparison of Confocal Laser Endomicroscopic IN Vivo Diagnosis and EX Vivo Examination (INDEX Study) Against Surgical Histopathology of Cystic Pancreatic Lesions
Brief Title: Comparison of CLE in Vivo Diagnosis and ex Vivo Examination Against Surgical Histopathology of CPL
Acronym: INDEX
Status: Completed | Type: Observational
Sponsor: Somashekar Krishna (Other)
Responsible Party: Sponsor-Investigator, Somashekar Krishna, Assistant Professor-Clinical, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2014C0205
Record Dates: First submitted 2015-07-30; First posted 2015-08-06 (Estimated); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Cystic Pancreatic Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: None Retained — Fluid from cyst in pancreas
Oversight: Data Monitoring Committee: No

SUMMARY:
Comparison of confocal laser endomicroscopic in vivo diagnosis and ex vivo examination against surgical histopathology of cystic pancreatic lesions.

DETAILED DESCRIPTION:
The primary objective of the study is to assess the ability of nCLE (AQ-Flex) to accurately diagnose the type of CPL by comparing in vivo and ex vivo CLE patterns to final histopathology of surgically resected CPLs. The primary endpoints are whether or not the CLE diagnosis correlates with final diagnosis (yes vs. no).

ELIGIBILITY:
Inclusion Criteria:

For in vivo nCLE (needle-based confocal laser endomicroscopy) (Part 1):

* Patient age 18 years and older
* All patients referred for EUS-FNA (endoscopic ultrasound - fine needle aspiration) of accessible CPL (cystic pancreatic lesion)
* The minimum size of the cyst should be ≥ 1.5 cm as determined by prior cross-sectional imaging studies.

For ex vivo pCLE (probe-based confocal laser endomicroscopy) (Part 2):

* All patients must satisfy inclusive criteria for in vivo nCLE.
* All patients should have completed EUS-guided nCLE.
* All patients should have a CPL lesion referred for surgical removal based on recommended international consensus guidelines1 and inter-departmental consensus pancreatic tumor board meeting (departments of surgical oncology, radiology, pathology and gastroenterology).
* Patient participated and completed in vivo nCLE (Part 1)

Exclusion Criteria:

* Unable to obtain informed consent
* Unable to tolerate the procedure
* Women with known pregnancy at time of procedure
* Patient age less than 18 years
* Bleeding diathesis
* Lesion not accessible by EUS guided FNA
* Allergy to fluorescein.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Cystic Pancreatic Lesions
Sampling Method: Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Diagnosis of cystic pancreatic lesion (CPL) using nCLE (confocal laser endomicroscopy) | 12 months
  Comparing the ability of nCLE to accurately diagnose the type of CPL by comparing in vivo and ex vivo CLE patterns to final histopathology of surgically resected CPLs.

SECONDARY OUTCOMES:
Detection of high-grade dysplasia and/or adenocarcinoma by CLE imaging | 12 months
CLE imaging interpretation variation | 12 months
  Calculate inter-observer variation in CLE image interpretation

CONTACTS AND LOCATIONS:
Overall Officials: Somashekar Krishna, MD, MPH, Principal Investigator — Ohio State Wexner Medical Center
Locations (1):
- OSU Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krishna SG, Hart PA, DeWitt JM, DiMaio CJ, Kongkam P, Napoleon B, Othman MO, Yew Tan DM, Strobel SG, Stanich PP, Patel A, Luthra AK, Chan MQ, Blaszczak AM, Lee D, El-Dika S, McCarthy ST, Walker JP, Arnold CA, Porter K, Conwell DL. EUS-guided confocal laser endomicroscopy: prediction of dysplasia in intraductal papillary mucinous neoplasms (with video). Gastrointest Endosc. 2020 Mar;91(3):551-563.e5. doi: 10.1016/j.gie.2019.09.014. Epub 2019 Sep 19. PMID 31542380
- [Derived] Krishna SG, Hart PA, Malli A, Kruger AJ, McCarthy ST, El-Dika S, Walker JP, Dillhoff ME, Manilchuk A, Schmidt CR, Pawlik TM, Porter K, Arnold CA, Cruz-Monserrate Z, Conwell DL. Endoscopic Ultrasound-Guided Confocal Laser Endomicroscopy Increases Accuracy of Differentiation of Pancreatic Cystic Lesions. Clin Gastroenterol Hepatol. 2020 Feb;18(2):432-440.e6. doi: 10.1016/j.cgh.2019.06.010. Epub 2019 Jun 18. PMID 31220640
- [Derived] Krishna SG, Brugge WR, Dewitt JM, Kongkam P, Napoleon B, Robles-Medranda C, Tan D, El-Dika S, McCarthy S, Walker J, Dillhoff ME, Manilchuk A, Schmidt C, Swanson B, Shah ZK, Hart PA, Conwell DL. Needle-based confocal laser endomicroscopy for the diagnosis of pancreatic cystic lesions: an international external interobserver and intraobserver study (with videos). Gastrointest Endosc. 2017 Oct;86(4):644-654.e2. doi: 10.1016/j.gie.2017.03.002. Epub 2017 Mar 10. PMID 28286093
- [Derived] Krishna SG, Swanson B, Hart PA, El-Dika S, Walker JP, McCarthy ST, Malli A, Shah ZK, Conwell DL. Validation of diagnostic characteristics of needle based confocal laser endomicroscopy in differentiation of pancreatic cystic lesions. Endosc Int Open. 2016 Nov;4(11):E1124-E1135. doi: 10.1055/s-0042-116491. Epub 2016 Sep 30. PMID 27853737